CLINICAL TRIAL: NCT05460624
Title: Daily Egg Consumption and Cognitive Function in Older Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study funding terminated prior to recruitment
Sponsor: Indiana University (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Andrew Brown, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13618
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Cognition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be conducted before randomization at baseline and by individuals blinded to the treatment assignments at follow-up. Data will be analyzed prior to unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants randomized to the intervention group will receive six premade egg-containing breakfast meals per week in the form of a 3-day rotating menu. Each meal contains 2 eggs to provide 12 eggs per week for a duration of 12 weeks.
  Interventions: Other: Egg-containing breakfast
- Control group (Other): Participants randomized to the control group will receive breakfast meals in the form of a 3-day rotating menu including typical foods found in American diets excluding eggs, e.g., corn flakes, milk, sausage, granola bars, fruit. Control recipes are matched to the intervention foods on total energy and saturated fat and to the 'What We Eat in America' on percent energy from macronutrients.
  Interventions: Other: Typical American-style breakfast excluding eggs

INTERVENTIONS:
Other: Egg-containing breakfast — Involves participants eating six premade egg-containing breakfast meals per week for 12 weeks. Each meal contains 2 eggs to provide 12 eggs per week.
  Arms: Intervention group
Other: Typical American-style breakfast excluding eggs — Involves participants eating six premade egg-excluding breakfast meals per week for 12 weeks. Breakfast meals are matched to the intervention egg-containing breakfast meals on total energy and saturated fat and to the 'What We Eat in America' on percent energy from macronutrients.
  Arms: Control group

SUMMARY:
The purpose of this study is to test the effects of provisioning twelve eggs weekly, incorporated into breakfast meals, on composite scores of executive functioning and memory using the CNSVS computerized test platform in older adults in a randomized study.

DETAILED DESCRIPTION:
Procedure: This study will test the effects of incorporating eggs at breakfast versus breakfasts that match a typical American breakfast on executive function and composite memory in adults 65 to 90 years old.

Randomization: Participants will be randomized using a permuted block randomization scheme to balance randomization across time with rolling enrollment, while ensuring allocation concealment through block sizes unknown to the investigators. Randomization will be also stratified by whether the individual participant is being randomized or multiple people from the same household (e.g., a couple being randomized together). This is to balance the number of randomized individual participants and households across the two conditions. Participants will be assigned sequentially

Analysis plan: An intention-to-treat analysis approach will be followed for data analysis. Primary statistical approach will be linear mixed models, including time, group, and their interaction as factors, where the interaction is the main test of interest to determine if the treatment group improved significantly more than the control group. The model will also include random effects for subjects (to account for repeated measurements) and for households (to adjust for clustering effect). Covariates for pre-randomization variables such as age, sex, education level, and computer familiarity may be included to account for variation in the outcomes and thereby improve power for the test of the intervention. For joint primary outcomes, we will split alpha of 0.05 between the two outcomes (p<0.025 for two-sided statistical significance). We will perform a compliers (threshold to be specified) and completers (those with both pre- and post-values) analysis as pre-specific secondary analyses on the primary outcomes. For pre-specified secondary outcomes, we will use the primary approach for the list of secondary outcomes. Results will be presented with and without multiple comparison or false discovery rate (FDR) corrections, and all analyzed outcomes will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Participant has autonomy over their food choices.
* Participant has the common appliances for storing refrigerated and frozen foods (i.e., refrigerator and freezer).
* Participant has common appliances to defrost/prepare foods (e.g., microwave oven, oven, stove, etc.).
* Participant has sufficient corrected visual acuity to read simple instructions on a computer/laptop screen
* Participant has a CNSVS standard (age-matched) score of 85-105 (inclusive) for either the domain composite memory (raw score is the sum of verbal memory score and visual memory score) or the domain executive function, and 80-110 for the other.
* Participant has no plans to change their routine (physical activity pattern, dietary habits, sleep pattern, smoking habits) during the study period unless advised as part of study participation.
* Participant is willing to follow screening/assessment visit instructions.
* Participant is willing to consume the study foods as provided at the breakfast meals during the study period.
* Participant is willing and able to visit IUB campus on specified in-person visit days.
* Participant understands the study procedures and signs the informed consent to participate in the study and is willing to complete study procedures.

Exclusion Criteria:

* Participant is not fully vaccinated for COVID-19.
* Participant reports habitually consuming greater than 5.5 eggs per week.
* Participant has sensitivity, allergy, taste aversion, or other aversion (e.g., vegan) to any ingredient of the study food.
* Participant has substantial dietary restrictions (e.g., chronic kidney disease or familial hypercholesterolemia diet) that, based on the judgment of the Principal Investigator, would interfere with the intervention.
* Participant has an established diagnosis of or is under treatment for dementia or ADHD. Anxiety or depression are not exclusionary.
* Participant is under active chemotherapy treatment.
* Participant is participating in a parallel research study that, based on the judgment of the Principal Investigator, would interfere with his or her ability to comply with the study protocol, or which might confound the interpretation of the study results.
* Participant is not able to read.
* Participant reports current use of cognitive enhancing medications, attention/concentration enhancing medications, anticonvulsant medications, and mood stabilizing medications.
* Participant has a condition that, based on the judgment of the Principal Investigator, would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Composite Memory | 12-week
  Derived from the CNSVS verbal and visual memory test scores
Executive Function | 12-week
  Derived from Shifting Attention Test (SAT) from CNSVS battery of tests

SECONDARY OUTCOMES:
Verbal memory | 12-week
  Derived from verbal memory test of CNSVS battery of tests
Visual memory | 12-week
  Derived from visual memory test of CNSVS battery of tests
Processing speed | 12-week
  Derived from symbol digit coding test of CNSVS battery of tests
Reaction time | 12-week
  Derived from Stroop test of CNSVS battery of tests
Simple Attention | 12-week
  Derived from continuous performance of CNSVS battery of tests
Working memory | 12-week
  Derived from 4-Part continuous performance of CNSVS battery of tests
Sustained Attention | 12-week
  Derived from 4-Part continuous performance of CNSVS battery of tests

OTHER OUTCOMES:
Dietary intakes | 12-week
  Measurement tool: 3-day food record
Physical performance | 12-week
  Measurement tool: The Short Physical Performance Battery (SPPB)
Serum total cholesterol | 12-week
Serum LDL cholesterol | 12-week
Serum HDL cholesterol | 12-week
Serum total triglycerides | 12-week
Blood Pressure | 12-week
Heart rate | 12-week
Skin carotenoids score | 12-week
  Measurement tool: The Vegie Meter®
Body composition | 12-week
  Measurement tool: Dual-energy X-ray absorptiometry (DEXA)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Brown, PhD, Principal Investigator — Indiana University, Bloomington
Locations (1):
- Indiana University-Bloomington, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All deidentified data and statistical code used for publication of the study results will be accessible publicly for other researchers to be able to reproduce and/or verify published results after confirmation that deidentified data cannot be reasonably statistically re-identified.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately
Access Criteria: Publicly available to anyone for the purpose of reproducing and/or verifying published results.